CLINICAL TRIAL: NCT03363360
Title: Comprehensive Awareness and Control in Diabetes Patients in China Jiangxi: A Cross-Sectional Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, YunFeng Shen, professor, Second Affiliated Hospital of Nanchang University
Other Study IDs: DM20161201
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: To Assess the Level of Control of Blood Glucose, Blood Pressure, and Blood Lipids Among Patients With Type 2 Diabetes in Jiangxi Province

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a multicenter, sub-center contrast, cross-sectional survey.The primary objective of this study was to assess the Comprehensive Awareness and Control of blood glucose, blood pressure, and blood lipids among patients with type 2 diabetes in China Jiangxi. An additional objective was to investigate the impact of hospital type on clinical outcomes.

DETAILED DESCRIPTION:
Background: With the continuous improvement of living standards in the past 30 years, the lifestyle and diet of Chinese people have undergone significant changes, leading to a significant increase in the prevalence of diabetes, hypertension and lipid metabolism disorders. Prevention and control work is also increasingly valued. At present, there is no research on the awareness rates and control rates of blood glucose, blood pressure and blood lipids in diabetic patients in Jiangxi Province. During the 13th Five-Year Plan period, the country has vigorously promoted the grading system of chronic non-communicable diseases, but there is a big gap between the levels of disease management in different levels of hospitals.

Methods:The province's multi-center, sub-center control, cross-sectional survey, the number of cases planned to be included in 10000 cases. Patient Access: Within 2 years from the date of the study (December 2016), eligible patients were screened out of outpatients in the participating hospitals, and patients were reviewed and informed of the informed consent.Inclusion criteria: in line with the WHO1999 diabetes diagnostic criteria; age 20-80 years; duration of 1 year or more; signed informed consent. Exclusion criteria: at the same time using other experimental drugs or in other clinical trials; gestational diabetes, other special types of diabetes; in acute infection, trauma and other stress conditions and the acute phase of the disease and other anomalies; patients with malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years to 80 years who were diagnosed with diabetes according to the World Health Organization criteria, at least 1 years before screening,written informed consent

Exclusion Criteria:

* Patients if they were pregnant or Other special types of diabetes, Patients with malignant tumor,participating in any other clinical studies, In phase of acute infection, trauma, such as stress state and acute phase of disease and other anomalies

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 to 80 - year - old diabetic patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | The first 30 days or seven days after the visit
  HbA1c <7%
TC | The first 30 days or seven days after the visit
  TC<5.2mmol/L
TG | The first 30 days or seven days after the visit
  TG<1.7mmol/L
LDL-C | The first 30 days or seven days after the visit
  LDL-C<3.3mmol/L
HDL-C | The first 30 days or seven days after the visit
  HDL-C>1.0mmol/L

SECONDARY OUTCOMES:
blood pressure | On the day of the visit
  systolic blood pressure <130 mm Hg, diastolic blood pressure <80 mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- No.1MinDeRoad, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes
In the form of a paper published based on the results of the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 1 years of completion of the study
Access Criteria: Researchers who need the results of this study